CLINICAL TRIAL: NCT04713241
Title: A Feasibility Study of Acupuncture for the Treatment of Postoperative Ileus After Gastrointestinal Surgery
Brief Title: Acupuncture for the Treatment of Postoperative Ileus After Gastrointestinal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3220
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Ileus; Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: SOC (Active Comparator): Participants will receive the SOC and will also be asked to complete questionnaires to rate their symptoms
  Interventions: Other: Standard of Care Bowel rest
- Group B: Electro-Acupuncture (Experimental): Participants will receive the SOC + a daily 20-30 minute electro-acupuncture treatment from the time of randomization until the return of bowel function. The first treatment will be provided within 48 hours after the diagnosis of postoperative ileus. Participants will receive acupuncture every day until normal bowel movement function returns.
  Interventions: Procedure: Electro-acupuncture; Other: Standard of Care Bowel rest

INTERVENTIONS:
Procedure: Electro-acupuncture — 20-30 minute acupuncture treatment in sessions from start of study (within 48 hours of diagnosis) to return of bowel functions
  A practitioner stimulates certain points on the body by placing thin needles in the skin. Electrical stimulation is then added to some of the needles. This involves placing wires on the needles, which are connected to a machine that delivers a weak electrical current through the wires. The strength of the electrical current will be changed slowly until it is at a comfortable level.
  Arms: Group B: Electro-Acupuncture
Other: Standard of Care Bowel rest — Bowel rest with NPO status and placement of nasogastric tube (NGT) if clinically indicated

SUMMARY:
The goal of this study is to learn if electro-acupuncture is a feasible treatment option for postoperative ileus after abdominal surgery. The second goal of this study is to evaluate the time to resolution of postoperative ileus after receiving electro-acupuncture treatments.

DETAILED DESCRIPTION:
Postoperative ileus is one of the most common complications following abdominal surgery. Despite significant advances in prevention, postoperative ileus continues to be a clinical issue. For patients experiencing postoperative ileus after a bowel resection, current treatment includes bowel rest, reduction of oral diet, and possible nasogastric tube placement while waiting for the postoperative ileus to resolve. Postoperative ileus results in postoperative complications, discomfort, and increases hospital stay. Electro-acupuncture treatment could potentially expedite the return of bowel function, reducing length of stay and increasing comfort. Additionally, acupuncture has been shown to be helpful for pain and nausea management, and thus may reduce the need for opioid and anti-nausea medications.

This study includes two groups. Both groups will be treated with conservative standard care (SOC), including bowel rest with nothing by mouth (NPO) status and placement of nasogastric tube if clinically necessary. Participants in both groups will continue on SOC postoperative recovery care with early feeding and ambulation, along with minimizing opioid use.

Group A: Participants assigned to group A will receive the SOC treatment described above and will also be asked to complete questionnaires to rate their symptoms.

Group B: Participants assigned to group B will receive the SOC described above and be given a daily 20-30 minute acupuncture treatment from the time of randomization until the return

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent document, and be willing to follow protocol requirements
* Diagnosis of gastrointestinal cancer
* Bowel resection was performed via an open or laparoscopic approach
* Diagnosis of POI defined as one or more of the following criteria: 1) return to NPO status after initial attempts at oral diet, and/or 2) need for placement of nasogastric tube after surgery.
* Willingness to comply with all study interventions of acupuncture

Exclusion Criteria:

* Active Infection at or near the acupuncture site or systemic infection (e.g. sepsis)
* Physical deformities that could interfere with accurate acupuncture and point location
* Concurrent use of other alternative medicines such as herbal agents and high dose vitamins and minerals
* Known coagulopathy or taking heparin (including low molecular weight heparin) at full anti-coagulation doses (prophylaxis is allowed) or Coumadin at any dose. Patients on aspirin or non-steroidal anti-inflammatories or other antiplatelet medicines will be allowed to participate
* Platelets <50 H K/UL in the past 30 days
* White Blood Cells (WBCs) <3.0 K/UL or Absolute Neutrophil Count (ANC) <1500 K/UL in the past 30 days
* INR >5 in the past 30 days
* Liver failure defined as liver function test >5x upper limit of normal
* Implanted electrical device such as a cardiac pacemaker, insulin pump or pain pump
* Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry
* Previous acupuncture treatment for any indications within 30 days of enrollment
* Currently pregnant
* Grade III lymphedema/lymphedema considered severe by the treating clinician
* Chronic daily opioid use prior to admission
* Enrollment in another surgical clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by acceptance rate of participation in study | An average of 1 day post-treatment
  Feasibility of acupuncture in study group as measured by acceptance rate of participation in study. Acceptance rate greater than 50% of patients being willing to participate will be considered feasible

SECONDARY OUTCOMES:
Time of ability to tolerate oral diet (liquid and solid food in hours) | An average of 1 day post-treatment
  Time to resolution of Postoperative ileus (POI) as measured by time of ability to tolerate oral diet (liquid and solid food in hours)
  Reported in mean, standard deviation as well as the five number summary including the 25th, 50th, and 75th percentiles, the minimum and maximum values
Nasogastric tube (NG TB) output | An average of 1 day post-treatment
  NG tube output, defined as volume of fluid collected from the NG TB
  Reported in mean, standard deviation as well as the five number summary including the 25th, 50th, and 75th percentiles, the minimum and maximum values

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request to members of the general public and scientific community at the conclusion and publication of the study results